CLINICAL TRIAL: NCT00503152
Title: A Prospective, Randomized, Probe Trial to Evaluate Whether, at Comparable Blood Pressure Control, Combined Therapy With the ACEI Benazepril and the ARB Valsartan, Reduces the Incidence of Microalbuminuria More Effectively Than BEN or VAL Alone in Hypertensive Patients With Type 2 Diabetes and High-normal Albuminuria
Brief Title: Preventing Microalbuminuria in Type 2 Diabetes
Acronym: VARIETY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Agenzia Italiana del Farmaco (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VARIETY; 2006-005954-62 (EudraCT Number)
Record Dates: First submitted 2007-07-17; First posted 2007-07-18 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — benazepril; Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- benazepril (Experimental)
  Interventions: Drug: Benazepril
- valsartan (Experimental)
  Interventions: Drug: Valsartan
- benazepril/valsartan (Experimental)
  Interventions: Drug: Benazepril/Valsartan

INTERVENTIONS:
Drug: Benazepril — After one month wash-out from previous RAS (ARB or ACE) inhibitor therapy, patients satisfying the inclusion/exclusion criteria will be randomly given equivalent doses (half the standard doses recommended by the manufacturer for blood pressure control) of benazepril (10 mg/day) or valsartan (160 mg/day) or one fourth of the standard doses of both agents in combination (benazepril 5 mg/day and valsartan 80 mg/day). If well tolerated, treatment will be up-titrated to full dose of benazepril (20 mg/day) or valsartan (320 mg/day) or one half of the standard doses of both agents in combination (benazepril 10 mg/day and valsartan 160 mg/day).
  Arms: benazepril
Drug: Valsartan — After one month wash-out from previous RAS (ARB or ACE) inhibitor therapy, patients satisfying the inclusion/exclusion criteria will be randomly given equivalent doses (half the standard doses recommended by the manufacturer for blood pressure control) of benazepril (10 mg/day) or valsartan (160 mg/day) or one fourth of the standard doses of both agents in combination (benazepril 5 mg/day and valsartan 80 mg/day). If well tolerated, treatment will be up-titrated to full dose of benazepril (20 mg/day) or valsartan (320 mg/day) or one half of the standard doses of both agents in combination (benazepril 10 mg/day and valsartan 160 mg/day).
  Arms: valsartan
Drug: Benazepril/Valsartan — After one month wash-out from previous RAS (ARB or ACE) inhibitor therapy, patients satisfying the inclusion/exclusion criteria will be randomly given equivalent doses (half the standard doses recommended by the manufacturer for blood pressure control) of benazepril (10 mg/day) or valsartan (160 mg/day) or one fourth of the standard doses of both agents in combination (benazepril 5 mg/day and valsartan 80 mg/day). If well tolerated, treatment will be up-titrated to full dose of benazepril (20 mg/day) or valsartan (320 mg/day) or one half of the standard doses of both agents in combination (benazepril 10 mg/day and valsartan 160 mg/day).
  Arms: benazepril/valsartan

SUMMARY:
In people with type 2 diabetes, microalbuminuria is a strong, independent risk factor for diabetic nephropathy and cardiovascular morbidity and mortality. ACE inhibitor therapy decreased the risk of microalbuminuria in hypertensive subjects with type 2 diabetes and normoalbuminuria by about 40%. Available data suggest that angiotensin II receptor blockers (ARBs) might have a similar renoprotective effect and that this effect might be increased by combined ACE inhibitor therapy.

The study will evaluate the effects, at similar blood pressure control (systolic/diastolic <130/80 mmHg), for a period of three years, of dual renin-angiotensin-system (RAS) blockade by benazepril and valsartan combination therapy as compared to single RAS blockade by benazepril or valsartan alone on microalbuminuria and cardiovascular events in high-risk patients with type 2 diabetes, creatinine <1.5 mg/dl, no evidence of microalbuminuria but at high risk of renal disease, with hypertension and a urinary albumin excretion between 7 and 19 microgram/min. The relationship between albuminuria and cardiovascular outcomes will also be evaluated.

The study is expected to show a more effective prevention of microalbuminuria and cardiovascular events with combined than with single drug ACE inhibitor or ARB therapy. As compared to ACE inhibitor, ARB therapy is expected to have a similar effect on microalbuminuria, but an inferior cardioprotective effect. Applied to clinical practice, the findings should help preventing renal and cardiovascular complications, and related treatment costs, of type 2 diabetes.

DETAILED DESCRIPTION:
Nephropathy of type 2 diabetes is the leading cause of end stage renal disease (ESRD) in the world.According to the World Health Organization (WHO), diabetes affects over 170 million people, and, due to progressive aging of the population, life-style modifications and increasing burden of obesity, this number is expected to rise to 370 millions by 2030. About one third of those affected will eventually have progressive deterioration of renal function Untreated, these patients progress to ESRD within 10 years or die prematurely because of cardiovascular complications (that are 10-fold more frequent in diabetics with nephropathy than in those without and the general population). Costs for renal replacement therapy of these patients - and for treatment of related complications - are also progressively increasing.

Persistent microalbuminuria is the first clinical sign of renal dysfunction in diabetic patients and progresses to overt proteinuria in 20 to 40 percent of cases. In 10 to 50 percent of patients with proteinuria, chronic kidney disease develops that ultimately requires dialysis or transplantation. Of great concern, 40 to 50 percent of type 2 diabetic patients with microalbuminuria eventually die of cardiovascular disease.Thus, preventing (or delaying) the development of microalbuminuria is a key treatment goal for renoprotection and, possibly, for cardioprotection.

A large scale randomized trial, the BErgamo NEphrologic DIabetes Complications Trial (BENEDICT) found that treatment with the ACE-inhibitor trandolapril (either alone or combined to the calcium channel blocker verapamil) significantly reduced the incidence of microalbuminuria in 1204 patients with type 2 diabetes and hypertension, but normal urinary albumin excretion, as compared with placebo. The effect of preventing microalbuminuria exceeded expectations based on changes in blood pressure alone and was not enhanced by combined calcium channel blocker therapy.

Studies in patients with type 2 diabetes and micro- or macro- albuminuria clearly show that ARBs can have renoprotective effect but trials evaluating the effects of angiotensin receptor blockers (ARBs) on the incidence of microalbuminuria in type 2 diabetic patients with normal urinary albumin excretion rate are missing.

Whether the beneficial effect against the development of microalbuminuria is enhanced when ACE inhibitors and ARBs are given in combination is not established so far. However, finding that combined ACE inhibitor and ARB therapy more effectively than single drug RAS blockade reduced albuminuria or proteinuria in subjects with type 2 diabetes and slowed progression to ESRD in those with non-diabetic chronic nephropathies, suggests that the renoprotective effect of combined therapy could be superior to that of single drug blockade of the RAS also in diabetic patients with no evidence of renal disease.

Post hoc analyses of the BENEDICT trial found that high-normal albuminuria at baseline evaluation (defined as a urinary albumin excretion rate between 10 µg/min and the upper limit for study entry: 19 µg/min) was the strongest baseline predictor of subsequent development of microalbuminuria. Indeed, regardless of treatment randomization, 69 of 271 (25.5%) patients with high-normal albuminuria (urinary albumin excretion >10µg/min) progressed to the end point as compared to only 32 of 933 (3.4%) with low-normal albuminuria (<10%). Thus, large-part of the excess risk for microalbuminuria observed in people with type 2 diabetes is associated with high-normal albuminuria.

In addition, this clinical trial might have a clinical relevance for the Italian National Health service (SSN): applied to clinical practice the results should help in reducing renal and cardiovascular complications and related treatment costs, of type 2 diabetes.

Aims Primary To evaluate whether, at comparable blood pressure control, dual RAS blockade with combined therapy with halved doses of benazepril (10 mg/day) and valsartan (160 mg/day) reduces the incidence of microalbuminuria more effectively than single drug RAS blockade by full doses of benazepril (20 mg/day) given alone in high-risk patients with type 2 diabetes, hypertension and high normal albuminuria.

Secondary

* To evaluate whether, at comparable blood pressure control, dual RAS blockade with combined therapy with halved doses of benazepril (10 mg/day) and valsartan (160 mg/day) reduces the incidence of microalbuminuria more effectively than valsartan (320 mg/day) given alone in high-risk patients with type 2 diabetes, hypertension and high normal albuminuria.
* To evaluate whether, at comparable blood pressure control, the effects of benazepril and valsartan therapy are similar or whether, alternatively, one of the two treatments offer a superior protective effect against the development of microalbuminuria in the above study population.
* To evaluate the effects of the three study treatments on the incidence of fatal and non-fatal cardiovascular events, regression to low-normal albuminuria (urinary albumin excretion <7 µg/min), albuminuria (considered as a continuous variable), serum creatinine, lipid profile, and GFR (in a representative subgroup);
* To assess the relationships, in the study group as a whole and within each treatment group, between renal outcome variables (including microalbuminuria and time-dependent changes in albuminuria) and fatal and non-fatal cardiovascular events, between achieved blood pressure or metabolic control and renal and/or cardiovascular outcome variables and between achieved albuminuria reduction or residual follow-up albuminuria and renal and/or cardiovascular outcome variables.

Design This will be a multicenter, Prospective, Randomized, Open label, Blinded End point (PROBE) trial of 3-year treatment with halved doses of benazepril (10 mg/day) and valsartan (160 mg/day) given in combination, or full doses of both benazepril (20 mg/day), or valsartan (320 mg/day) given alone in 1020 consenting patients >40 year old, with type 2 diabetes (WHO criteria), serum creatinine <1.5 mg/dl, high-normal albuminuria (UAE >7 and <20 µg/min in at least 2 of 3 overnight urine collections), and no specific contraindications to the study drugs. Primary outcome variable will be microalbuminuria (UAE > 20µg /min in at least 2 of 3 overnight urine collections in two consecutive visits 2 months apart) and primary comparison will be between the combined benazepril plus valsartan and the benazepril alone groups. The analysis will have an 80% power to detect (p=0.05, two-side test) a 40% difference in the incidence of microalbuminuria.

ELIGIBILITY:
Inclusion Criteria:

* Males and females >40 years old;
* High-risk subjects with type 2 diabetes (WHO criteria);
* History of diabetes not exceeding 25 years;
* High blood pressure (systolic and/or diastolic blood pressure >135/85 mmHg or concomitant treatment with blood pressure lowering medications);
* Serum creatinine concentration <1.5 mg/dl;
* Overnight urinary albumin excretion (in at least 2 of 3 consecutive overnight urine collections) ≥ 7 and <20 µg/min;
* Legal capacity;
* Written informed consent.

Exclusion Criteria:

* Uncontrolled diabetes (glycated hemoglobin >11%);
* Specific contraindications or history of hypersensitivity to the study drugs;
* Serum potassium ≥ 5.5 mEq/L despite diuretic therapy, and optimized metabolic and acid/base control;
* Bilateral renal artery stenosis;
* Previous history of allergy or intolerance, or evidence of immunologically-mediated renal disease, systemic diseases, cancer;
* Drug or alcohol abuse;
* Any chronic clinical conditions that may affect completion of the trial or confound data interpretation;
* Pregnancy or lactating;
* Women of childbearing potential without following a scientifically accepted form of contraception;
* Legal incapacity and/or other circumstances rendering the patient unable to understand the nature, scope and possible consequence of the trial;
* Evidence of an uncooperative attitude;
* Any evidence that patient will not be able to complete the trial follow-up.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 612 (Actual)
Dates: Start 2007-05; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Development of persistent microalbuminuria (i.e. urinary albumin excretion rate >20 µg/min in at least 2 of 3 consecutive overnight urine collections confirmed in two consecutive visits). Whenever a patient will be found to have 2 of 3 collections in the | 2 times a year

SECONDARY OUTCOMES:
Regression to low-normal albuminuria (i.e. urinary albumin excretion rate <7 µg/min in at least 2 of 3 consecutive overnight urine collections confirmed in two consecutive visits); Albuminuria (considered as a continuous variable); Serum creatinine (v | 2 times a year

CONTACTS AND LOCATIONS:
Overall Officials: Piero Ruggenenti, MD, Study Director — Mario Negri Institute for Pharmacological Research
Locations (9):
- Italy (9):
  - Hospital "Azienda Ospedaliera di Treviglio e Caravaggio" - Diabetologic Ambulatory of Ponte San Pietro, Ponte San Pietro, Bergamo
  - Clinical Research Center for Rare Diseases "Aldo e Cele Daccò", Ranica, Bergamo
  - Hospital "Azienda Ospedaliera di Treviglio e Caravaggio" Unit of Diabetology and Metabolic Diseases, Romano di Lombardia, Bergamo
  - Hospital "Bolognini", Seriate, Bergamo
  - Hospital "Azienda Ospedaliera di Treviglio-Caravaggio"Unit of Diabetology and Metabolic Diseases, Treviglio, Bergamo
  - Hospital "Casa Sollievo della Sofferenza" - Division of Endocrinology, San Giovanni Rotondo, Foggia
  - Hospital "Azienda Ospedaliera Ospedali Riuniti di Bergamo" - Unit of Diabetology, Bergamo
  - IRCCS San Raffaele - Unit of General Medicine, Milan
  - Azienda USL 2, Olbia

REFERENCES:
- [Derived] Ruggenenti P, Cortinovis M, Parvanova A, Trillini M, Iliev IP, Bossi AC, Belviso A, Aparicio MC, Trevisan R, Rota S, Perna A, Peracchi T, Rubis N, Martinetti D, Prandini S, Gaspari F, Carrara F, De Cosmo S, Tonolo G, Mangili R, Remuzzi G; VARIETY Study Organization. Preventing microalbuminuria with benazepril, valsartan, and benazepril-valsartan combination therapy in diabetic patients with high-normal albuminuria: A prospective, randomized, open-label, blinded endpoint (PROBE) study. PLoS Med. 2021 Jul 14;18(7):e1003691. doi: 10.1371/journal.pmed.1003691. eCollection 2021 Jul. PMID 34260595